CLINICAL TRIAL: NCT06061835
Title: Non-contrast Magnetic Resonance Angiography Efficacy and Safety Assessment for Perforators Mapping in Deep Inferior Epigastric Perforator Flap Breast Reconstruction
Brief Title: Non-contrast Magnetic Resonance Angiography in Deep Inferior Epigastric Perforator Flap Breast Reconstruction Planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MD05052023; Patent № RU 2023121330 (Other: Federal institute of industrial property)
Record Dates: First submitted 2023-09-16; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Postsurgical Acquired Absence of Organ
Keywords: Autologous breast reconstruction; Preoperative planning; Perforator mapping; Deep Inferior Epigastric Perforator Flap; Magnetic resonance angiography; Computed tomography angiography
MeSH Terms: conditions — Breast Neoplasms | interventions — diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-contrast MRA (MRA "-") (Experimental): Participants in this group underwent preoperative planning with a contrast-free magnetic resonance angiography (MRA) using an enhanced protocol that eliminates the use of potentially hazardous contrast agent and radiation exposure while providing high accuracy of visualization.
  Interventions: Other: Non-contrast MRA in preoperative perforator vessels mapping for deep inferior epigastric perforator (DIEP) flap breast reconstruction planning.
- CTA with contrast (CTA "+") (Other): Control group. Participants in this group underwent preoperative planning using the standard commonly used method - computed tomography angiography (CTA) with IV (intravenous) iodine-containing contrast injection.
  Interventions: Other: CTA with iodine contrast in preoperative perforator vessels mapping for deep inferior epigastric perforator (DIEP) flap breast reconstruction planning.

INTERVENTIONS:
Other: Non-contrast MRA in preoperative perforator vessels mapping for deep inferior epigastric perforator (DIEP) flap breast reconstruction planning. — Device: MRA scan Philips Ingenia 1.5 T (Royal Philips, Netherlands)
  Preprocedural patient's preparation: the study was performed on an empty stomach (at least 8 hours of fasting).
  Type of patient positioning. MRA scanning was performed in the prone position.
  Additional devices. The investigators placed the patient on her abdomen on a special coordinate system mesh, for the most precise and convenient way of marking.
  Scanning protocol. The investigators added T2 pulse sequence to increase the accuracy of muscle localization assessment and the point of vessel immersion into the muscle at TR and TE using a fat suppression program, wich allows receiving information from moving objects (including blood within the vascular lumen).
  Scan viewer program. OsiriX 10.0 Release
  Arms: Non-contrast MRA (MRA "-")
Other: CTA with iodine contrast in preoperative perforator vessels mapping for deep inferior epigastric perforator (DIEP) flap breast reconstruction planning. — Device: Device: Toshiba Aquilion 64 CTA scan machine (Toshiba Medical Systems, Tokyo, Japan).
  Preprocedural patient's preparation: A catheter was placed in the antecubital vein of one arm, and a bolus injection of 80 ml contrast medium (Omnipaque 300 mg/ml, GE Healthcare, Oslo, Norway, registration number P N015799/01 from July 31, 2003, international nonproprietary name is a Iohexol) was administered through a power injector (M. Schilling GmbH Medical Products, Germany) at 4 ml/s.
  Type of patient positioning. CTA scanning was performed in the supine position.
  Scan viewer program. OsiriX 10.0 Release
  Arms: CTA with contrast (CTA "+")

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of contrast-free magnetic resonance angiography (MRA) for deep inferior epigastric perforator flap planning. The investigators propose to perform a non-contrast MRA to achieve the following extremely important objectives: to avoid radiation exposure, minimize the risk of potentially harmful effects of contrast agents, and reduce the cost of the study.The investigators assume that the use of non-contrast MRA following our protocol including certain patient's positioning, a special pulse scanning sequence and perforators' projection method is effective and allows mapping of perforators without injecting a potential harmful contrast agent.

DETAILED DESCRIPTION:
Rationale. Contrast-free MRA is a new concept for preoperative planning in breast reconstruction that combines the advantages of magnetic resonance imaging (no ionising radiation exposure), requires no potentially harmful contrast agent, and at the same time is highly accurate.

Aim. The aim of the study is to evaluate the efficacy and safety of the contrast-free magnetic resonance angiography (MRA) for perforators mapping in deep inferior epigastric perforator flap planning.

Study design. A retro- and prospective non-randomised non-blinded cohort multicenter study is conducted at the at the Department of Plastic Surgery (Sechenov University, Moscow), and at the Department of Reconstructive and Plastic Surgery (Lancet Clinic, Moscow), with all patients recruited through a single surgical team and all imaging performed at a single institution.

Study population. The investigators plan to conduct a pilot phase of this study using non-contrast MRA in 100 patients and to compare imaging modalities used in deep inferior epigastric perforator flap breast reconstruction (computed tomography angiography with contrast, n=35 and non-contrast magnetic resonance angiography, n=100). Power analysis determine that no less than 35 patients in control group in this study considering 80 % power with 95 % significance. The first group (experimental, MRA "-" group) will be included patients who refused computed tomography angiography (CTA) with contrast due to a number of reasons such as fear of contrast agent administration, history of iodine allergy, fear of radiation exposure, etc was underwent MRA without contrast, and the second group (control, CTA "+" group) will be involved iodine-tolerance patients with healthy kidneys who underwent preoperative planning with a standard technique - CTA with IV iodine-containing contrast injection.

Interventions. Participants in first group (experimental, MRA "-" group) underwent preoperative planning with a contrast-free magnetic resonance angiography (MRA) using an improved contrast-free MRA protocol. MRA was performed on a magnetic resonance machine Philips Ingenia 1.5 T (Royal Philips, Netherlands). High accuracy is achieved by the following actions: certain preprocedural patient's preparation and positioning, special pulse scanning sequence and perforators projection method.

Preprocedural patient's preparation. The investigators added to the MRA protocol a requirement of performing the study on an empty stomach (at least 8 hours of fasting) in order to reduce gastrointestinal activity.

Modified type of patient positioning. The investigators suggest performing MRA scanning in the prone position in order to both limit abdominal wall movement (related to breathing, peristalsis, and aortic pulsation) and to provide the closest location of the target area (vessels) to the coil.

Furthermore, this move allowed to introduce a further trick that facilitated the surgeons' work at the marking stage: the investigators placed the patient on her abdomen on a 3D printed special mesh made of ABS (Acrylonitrile Butadiene Styrene) (the patent for invention № RU 2023118155). The mesh served as a coordinate system, crosshairs of which accommodate capsules with liquid (A), which allows obtaining on the image not only vessels but also all points of capsules to form a basic standardized mesh, coinciding on the image and on the patient's body that is necessary for the most precise and convenient way of marking.

Due to the image directly used for preoperative marking, the protocol of the MRA scans description was not used.

Special pulse sequence and additional series of MRA scans. MRA is performed on a magnetic resonance machine Philips Ingenia 1.5 T in the T2 pulse sequence (to increase the accuracy of muscle localization assessment and the point of vessel immersion into the muscle) at TR and TE using a fat-suppression program with no IV contrast injection, which allows receiving information from moving objects (including blood within the vascular lumen). The investigators have incorporated an additional series of T2 scans without fat suppression with high resolution (thickness of slices from 0.8 to 1.2 mm) and visualization of the muscle fibers, which allows us to determine the site where the vessels pierce the muscle, intramuscular course of the perforating vessels, and the topography of the area of interest with accurate determination of the perforating vessel relative to the anatomical landmarks.

Following scanning, the images were analysed by a plastic surgeon in the OsiriX 10.0 program. The main benefit of the images was extracted by creating multiplanar reconstructions (MPR) in Maximum Intensity Processing (MIP) mode. This mode allows the evaluation of the vessels in length, their lumen diameters and the study of their correlations and distances from each other for the purpose of target vessel selection.The MRA images required simultaneous evaluation in two planes: frontal and sagittal or frontal and axial. This allowed to the investigators to evaluate the localize the point of vessel immersion into the muscle, the extent and direction of the vessel in the muscle thickness and to localize the point of vessel penetration over the muscle with further direction of the vessel course and the point of communications between superficial and deep systems.

The second group participants (control, CTA "+"group) underwent the standard commonly used computed tomography angiography (CTA) IV (intravenous) iodine-containing contrast injection, and in the supine position. CTA was performed on a Toshiba Aquilion 64 CTA scan machine (Toshiba Medical Systems, Tokyo, Japan) according to the Research and Practical Center of Medical Radiology guidelines №12 from March 22, 2017.

Informed consent is obtained from each participant.

Main study parameters. The investigators plan to evaluate the results according to the following criteria: the concordance ratio, the overall operation time, the time of the pedicle cut, the length of the fascia incision, the intraoperative flap perfusion, the presence of early postoperative complications and their nature, the presence of emergent vascular revision surgery. In addition, the investigators plan to evaluate the following parameters: the flap ischemia time, the number of perforators included in the flap, the fact of superficial vein(s) inclusion in the flap, the length of the vascular pedicle.

ELIGIBILITY:
Inclusion Criteria:

* A female patients who underwent unilateral mastectomy due to breast cancer, in remission.
* At least 1 year after completion of radiotherapy.

Non-inclusion Criteria:

* A history of abdominal donor site free flaps or abdominoplasty.
* Inability to give consent.
* The expander with magnetic ports, claustrophobia, pregnancy and breastfeeding.
* Patients with severe hypertension, COPD, autoimmune disorders, SLE or poorly regulated diabetes
* The presence of psychiatric illness preventing participation in the study.

Exclusion Criteria:

* Patient's pregnancy diagnosed during the research period.
* Patient's refusal of surgery, patient's refusal of further participation in the study.
* The presence of concomitant diseases preventing participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients in both groups will be female.
Enrollment: 135 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The concordance ratio. | During the surgery.
  The investigators are use the information about each perforators' deviation (P1, P2, etc.) based on intraoperative finding (confirmation) and MRA or CTA data by more/less than 1 cm.
  Intraoperatively, the surgeon determined the distance from the umbilicus to the perforator vessel (by dropping a perpendicular line from umbilicus) and the distance from the point marked on the marking according to the MRA or CTA data to the found perforator vessel. Measurements performed using a 200 mm surgical ruler (Devemed, Germany).
The overall operation time (min). | Immediately after the surgery.
  The total operating time including downtime.
The time of the pedicle cut (min). | During the surgery.
  The investigators plan to evaluate the time of the pedicle cut from the beginning of surgery and from flap harvest, for the right and left vascular pedicle individually.
The length of the fascia incision (cm). | During the surgery.
  Intraoperatively, the surgeon measured the fascia incision length using a 200 mm surgical ruler (Devemed, Germany).
Intraoperative evaluation of flap perfusion. | During the surgery.
  The flap perfusion was assessed for capillary refill after the vascular pedicle clipping, after the vascular pedicle cutting, and at the end of the flap ischemia time (after the microvascular anastomosis formation) by applying mild pressure, using a hemostat handle. Pressure was then released and the flap observed for capillary refill. Refill was deemed positive if it occurred within 3 s.
Postoperative flap necrosis (%). | During the first week after surgery.
  The presence of flap necrosis was assessed during the first five days after surgery by evaluating capillary refill in thee flap and visually assessed the presence of the flap ischemia or necrosis as a percentage of the total flap.

SECONDARY OUTCOMES:
The flap ischemia time (min). | During the surgery.
  Flap ischemia time was assessed from the time of vascular pedicle cutoff to completion of microvascular anastomosis formation ( up to the beginning of blood flow).
The length of the vascular pedicle (cm). | During the surgery.
  After flap harvesting, the surgeon measured the vascular pedicle length using a 200 mm surgical ruler (Devemed, Germany).
The number of perforators included in the flap. | Immediately after the surgery.
  The investigators recorded the number of perforators included in the flap on each side of the flap.
Inclusion of superficial vein(s) in the flap. | Immediately after the surgery.
  The investigators recorded the fact of the superficial vein(s) inclusion in the flap, their number and localization (side of the flap).

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry V. Melnikov, MD, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University; Victor A. Gombolevskiy, MD, PhD, Principal Investigator — Artificial Intelligence Research Institute (AIRI)
Locations (2):
- Russia (2):
  - Lancet Clinic, Moscow
  - IMSechenovMMA, Moscow

IPD SHARING:
Plan to Share IPD: No
Due to the local ethics committee the investigators are unable to provide this data.